CLINICAL TRIAL: NCT06294847
Title: Ursodeoxycholic Acid (UDCA) as a Neuroprotective Adjuvant Treatment to Rhegmatogenous Retinal Detachment Surgery
Acronym: UDCA
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Hopital Foch (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2021_0025
Record Dates: First submitted 2024-02-28; First posted 2024-03-06 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Retinal Detachment
MeSH Terms: conditions — Retinal Detachment | interventions — Ursodeoxycholic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental arm: 'UDCA' (Experimental): Experimental arm: 'UDCA': Patients will be treated with ursodeoxycholic acid (UDCA), receiving a single dose of Ursolvan® (10mg/kg) orally within 24 hours before the surgical intervention, followed by a daily dose of 10mg/kg in two divided doses for 30 days.
  Interventions: Drug: Ursolvan
- Control arm: 'Placebo' (Placebo Comparator): Control arm: 'Placebo': Patients will receive a single dose of placebo orally within 24 hours before the surgical intervention, followed by two doses per day for 30 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ursolvan — single dose of Ursolvan® (10mg/kg) orally within 24 hours before the surgical intervention, followed by a daily dose of 10mg/kg in two divided doses for 30 days.
  Arms: Experimental arm: 'UDCA'
Drug: Placebo — Patients will receive a single dose of placebo orally within 24 hours before the surgical intervention, followed by two doses per day for 30 days
  Arms: Control arm: 'Placebo'

SUMMARY:
This study is indicated for patients with extended rhegmatogenous retinal detachment (RRD) (≥ 2 quadrants) with macula OFF lasting 7 days or less, pseudophakic or aphakic, and scheduled to undergo surgical intervention with vitrectomy and gas tamponade in one of the ophthalmology departments participating in the study.

The main objective is to assess the effectiveness of UDCA in visual acuity recovery at 3 months (i.e., the difference between preoperative visual acuity and visual acuity 3 months after surgery) in pseudophakic or aphakic patients who have undergone successful surgical intervention (reattachment of the retina) through vitrectomy and gas tamponade following rhegmatogenous retinal detachment (RRD).

120 patients will be enrolled and randomized in two groups:

* the experimental arm "UDCA Group," with oral administration of ursodeoxycholic acid (Ursolvan®)
* the control group "Placebo Group," with oral administration of the placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 years or older,
2. Scheduled to undergo surgical intervention through vitrectomy,
3. Aphakic or pseudophakic patients,
4. Experiencing rhegmatogenous retinal detachment affecting 2 quadrants or more,
5. Presenting with macula OFF (raised macula) for 7 days or less before the onset of symptoms,
6. Has signed a consent form,
7. Affiliated with a health insurance plan.

Exclusion Criteria:

1. Patients who have previously undergone vitrectomy for retinal detachment,
2. Patients with vitreous hemorrhage or any other associated retinal pathologies,
3. Monophthalmic patients,
4. Women of childbearing age without effective contraceptive methods,
5. Pregnant or lactating women,
6. Hypersensitivity to the active substance, bile acids, or any of the excipients in Ursolvan® (see §6.1.1 of this protocol),
7. Patients with peptic ulcers, acute or chronic liver disease, acute infection or inflammation of the gallbladder or bile ducts, recurrent gallstones, or obstruction of the bile ducts (common bile duct or cystic duct obstruction),
8. Patients with radiopaque calcified gallstones,
9. Patients with severe pancreatic disorders,
10. Patients with Crohn's disease, ulcerative colitis, or other intestinal diseases that may alter the enterohepatic circulation of bile acids,
11. Patients on oral treatment with cholestyramine, colestipol, antacids containing aluminum or magnesium hydroxide and/or smectite (aluminum oxide), cyclosporine, ciprofloxacin, nitrendipine, or dapsone,
12. Patients with galactose intolerance, Lapp lactase deficiency, or glucose and galactose malabsorption syndrome (rare hereditary diseases),
13. Patients participating or in the exclusion period following an interventional research with the use of prohibited medications in this study,
14. Patients under protective custody.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-08-20 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Difference in visual recovery (difference between preoperative and postoperative visual acuity) at 3 months postoperative (after a successful reapplication procedure) of at least 6 letters (ETDRS scale) between the two groups (treatment and placebo) | 3 months
  Difference in visual recovery (difference between preoperative and postoperative visual acuity) at 3 months postoperative (after a successful reapplication procedure) of at least 6 letters (Early Treatment Diabetic Retinopathy Study (ETDRS scale) between the two groups (treatment and placebo).
  The minimum and maximums valus :
  Minimum value is 6/95 equivalent in ETDRS letter score read at 4 m = 55. Maximum value is 6/6 equivalement in ETDRS letter score read at 4 m= 115. Higher score mean better ourcome

SECONDARY OUTCOMES:
Central Nervous Epithelium (CNE) thickness | 1, 3, and 6 months
  Central Nervous Epithelium (CNE) thickness, measured by SD-OCT (Spectral-Domain Optical Coherence Tomography), within the central 1mm compared to the contralateral eye in the treated group versus the placebo group (measurement adjusted to the contralateral eye to account for interindividual variability) at 1, 3, and 6 months.
Automated microperimetry at 1, 3, and 6 months: Macular sensitivity difference between the two groups. | 1, 3, and 6 months
  Automated microperimetry at 1, 3, and 6 months: Macular sensitivity difference between the two groups.
Contrast sensitivity measurement using the Clinic CSF2.0 application. | Day 7, Day 30, Day 60, Day 60, Day 90 and Day 180
  Contrast sensitivity measurement using the Clinic CSF2.012 application (Contrast sensitivity function 2.0 application).
Presence/absence of abnormal signs on optical coherence tomography (OCT) images (cysts, folds, membrane, ellipsoid zone, external limiting membrane). | 1, 3 and 6 months
  Presence/absence of abnormal signs on optical coherence tomography (OCT) images (cysts, folds, membrane, ellipsoid zone, external limiting membrane).
Retinal thickness measured by OCT (retinal layers and presence of cysts, layer segmentation and measurement in the central 1 and 3 mm in ETDRS quadrants). | 1, 3 and 6 months
  Retinal thickness measured by OCT (retinal layers and presence of cysts, layer segmentation and measurement in the central 1 and 3 mm in ETDRS quadrants).
Number of macular cones and retinal pigment epithelium (RPE) cells measured by Adaptive Optics at 1, 3, and 6 months with the "Cellularis" device that allows visualization of cones and RPE. | 1, 3 and 6 months
  Number of macular cones and retinal pigment epithelium (RPE) cells measured by Adaptive Optics at 1, 3, and 6 months with the "Cellularis" device that allows visualization of cones and RPE.
Blood test: liver parameters - AST (SGOT), ALT (SGPT), PAL, and γ-GT. | Day 7 and Day 30
  Blood test: liver parameters - AST (SGOT), ALT (SGPT), PAL, and γ-GT.
Evolution of the best visual acuity measured at Day 0, Day 7, Day 30, Day 60, Day 90, and Day 180: Difference between the treated and placebo groups in the progression curves of visual acuity. | Day 7 and Day 30
  Evolution of the best visual acuity measured at Day 0, Day 7, Day 30, Day 60, Day 90, and Day 180: Difference between the treated and placebo groups in the progression curves of visual acuity.
Presence of metamorphopsia. | 1, 3 and 6 months
  Presence of metamorphopsia.
Tolerance and occurrence of adverse events. | 1, 3 and 6 months
  Tolerance and occurrence of adverse events.
National Eye Institute Visual Functioning Questionnaire-25 (NEIVFQ-25) quality of life questionnaire before surgery, at ±7 days postoperative, and at 3 months postoperative. | 1, 3 and 6 months
  National Eye Institute Visual Functioning Questionnaire-25 (NEIVFQ-25) quality of life questionnaire before surgery, at ±7 days postoperative, and at 3 months postoperative.
Correlation between protein levels, bile acids, or other molecular markers in ocular and/or blood fluids and functional and anatomical ocular parameters pre- and post-operatively at different observation times. | 1 month
  Correlation between protein levels, bile acids, or other molecular markers in ocular and/or blood fluids and functional and anatomical ocular parameters pre- and post-operatively at different observation times.
Correlation between the effective duration of treatment and functional and anatomical outcomes at different observation times. | 6 months
  Correlation between the effective duration of treatment and functional and anatomical outcomes at different observation times.

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Hôpital Cochin, Paris
  - Hôpital Foch, Suresnes